CLINICAL TRIAL: NCT01752088
Title: Arthroscopic Repair of Subscapularis Tear :Clinical Results and MRI Analysis
Brief Title: Repair of Subscapularis Tear :Clinical Results and MRI Analysis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Lin Lin, Dr., Peking University Third Hospital
Other Study IDs: SSC2012
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Rupture Subscapularis Tendon
Keywords: apularis, MRI clinical, results

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to evaluate the magnetic resonance imaging (MRI) and clinical results of arthroscopic repair of subscapularis tears

DETAILED DESCRIPTION:
ROM UCLA Constant ASES VAS MRI Goutallier

ELIGIBILITY:
Inclusion Criteria:

- Patients suffering from rotator cuff injury scheduled for an arthroscopic procedure. A partial- or full-thickness subscapu-laris tendon tear

Exclusion Criteria:

- revision repairs or open repairs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from rotator cuff injury will be scheduled for an arthroscopic procedure
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical results and MRI analysis | 2 year
  ROM UCLA Constant ASES VAS MRI

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Denard PJ, Jiwani AZ, Ladermann A, Burkhart SS. Long-term outcome of a consecutive series of subscapularis tendon tears repaired arthroscopically. Arthroscopy. 2012 Nov;28(11):1587-91. doi: 10.1016/j.arthro.2012.02.031. Epub 2012 May 24. PMID 22632896